CLINICAL TRIAL: NCT03723785
Title: Investigation of Pharmacokinetics and Safety Profile of a Single Dose NNC0148-0287 C (Insulin 287) in Subjects With Various Degrees of Renal Impairment
Brief Title: A Research Study of How a New Medicine NNC0148-0287 C (Insulin 287) Works in the Body of People With Kidney Problems
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4226; 2017-004529-34 (EudraCT Number); U1111-1204-8972 (Other: World Health Organization)
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Participants with normal renal function (Experimental): Participants with normal renal function (glomerular filtration rate [GFR] of greater than or equal to 90 ml/min) will receive single dose of insulin 287 on Day 1.
  Interventions: Drug: Insulin icodec
- Participants with mildly decreased renal function (Experimental): Participants with mildly decreased renal function (GFR of 60 to less than 90 ml/min) will receive single dose of insulin 287 on Day 1.
  Interventions: Drug: Insulin icodec
- Participants with moderately decreased renal function (Experimental): Participants with moderately decreased renal function (GFR of 30 to less than 60 ml/min) will receive single dose of insulin 287 on Day 1.
  Interventions: Drug: Insulin icodec
- Participants with severely decreased renal function (Experimental): Participants with severely decreased renal function (GFR of less than 30 not requiring dialysis) will receive single dose of insulin 287 on Day 1.
  Interventions: Drug: Insulin icodec
- Participants with end-stage renal disease (Experimental): Participants with end-stage renal disease requiring haemodialysis will receive single dose of insulin 287 on Day 1.
  Interventions: Drug: Insulin icodec

INTERVENTIONS:
Drug: Insulin icodec — Participants will receive single dose of Insulin 287 subcutaneously (under the skin) on Day 1
  Other Names: Insulin 287

SUMMARY:
This study will be conducted to look at the effect of decreased kidney function when getting one dose of insulin 287 and to guide dosing recommendations in people who have altered kidney function. Insulin 287 works in the body for a long time (long-acting). It is taken once a day by injecting under the skin. The main target patient group for insulin 287 is people with type 2 diabetes. Participants will get just one injection. The study will last for up to 80 days. Participants will have 11 out-patient visits with the study doctor and one in-house visit of 3 days and 2 nights. Participants will have some assessments like several blood draws, electrocardiograms (ECGs), urine collections and capillary blood sugar tests. Participants cannot take part if they are hypersensitive to the study medicine, if they received any investigational product within 90 days before screening, or if they have certain diseases e.g. HIV or hepatitis or heart problems. Participants have to take photos if they experience any allergic reactions and send them to their study doctor. Participants' kidney function will be examined by a so called "Iohexol test".

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-75 years (both inclusive) at the time of signing informed consent.
* Body mass index between 18.5 and 32.0 kg/sqm (both inclusive).
* Meeting the pre-defined Glomerular Filtration Rate (GFR) values based on a measured GFR using an exogenous substance as tracer (renal group 1-4) or being in treatment with haemodialysis (renal group 5).

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product or related products.
* Impaired liver function defined as Alanine Aminotransferase (ALT) greater than or equal to 2.5 times or Bilirubin greater than 1.5 times upper limit of normal at screening.
* Drugs known to affect creatinine clearance including cephalosporin and aminoglycoside antibiotics, flucytosine, cisplatin, cimetidine and trimethoprim within 14 days or 5 half-lives prior to the day of dosing of IMP.
* Renal group 1 (healthy subjects) exclusively: Unwilling to avoid use of prescription medicinal products or non-prescription drugs, except routine use of vitamins, occasional use of paracetamol, topical medication and contraceptives, within 14 days prior to the day of dosing.
* Renal Group 2-5 (renal impairment) exclusively: 1) Any disorder, except for conditions associated with renal impairment in the groups of subjects with reduced renal function, which in the investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol. Subjects with heart failure of functional class III-IV according to New York Heart Association (NYHA), subjects with Chronic obstructive pulmonary disease (COPD) grade 4 according to Global Initiative on Obstructive Lung Disease (GOLD), subjects with asthma step 5 according to Global Initiative for Asthma (GINA), subjects diagnosed with diabetes, subjects with uncontrolled treated/untreated hypertension (systolic blood pressure greater than or equal to 180 mmHg and /or diastolic blood pressure greater than or equal to 100 mmHg assessed in supine position) and other co-morbidities in terminal stages or which are decompensated or unstable should not be included in the study. 2) Subject requiring haemodialysis treatment unable or unwilling to undergo haemodialysis scheduled according to the standard clinical regimen throughout the trial period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
AUCI287,0-840h,SD: Area under the serum insulin 287 concentration-time curve after a single dose | From 0 to 840 hours after trial product administration (visit 2 (study day 1))
  Measured in pmol*h/L

SECONDARY OUTCOMES:
Cmax,I287,SD: Maximum observed serum insulin 287 concentration after a single dose | From 0 to tz hours after trial product administration (visit 2 (study day 1)), where tz is the time of the last quantifiable concentration
  Measured in pmol/L
tmax,I287,SD: Time to maximum observed serum insulin 287 concentration after a single dose | From 0 to tz hours after trial product administration (visit 2 (study day 1)).
  Measured in hours
Number of adverse events | From trial product administration (visit 2 (study day 1)) until visit 13 (study day 43)
  Number of events
Change in anti-insulin 287 antibody level | From visit 2 (study day 1, pre-dose) to visit 13 (study day 43)
  Measured in % B/T (percentage of bound tracer measured after precipitation to total tracer)
Change in anti-insulin 287 antibody titres | From visit 2 (study day 1, pre-dose) to visit 13 (study day 43)
  Number of dilutions
Positive cross-reactive anti-human insulin antibodies | At visit 13 (study day 43)
  Number of patients with/without positive cross-reactive anti-human insulin antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Haahr H, Cieslarova B, Hingst JR, Jiang S, Kristensen NR, Kupcova V, Norgreen L, Wagner FH, Ignatenko S. The Effect of Various Degrees of Renal or Hepatic Impairment on the Pharmacokinetic Properties of Once-Weekly Insulin Icodec. Clin Pharmacokinet. 2024 Jun;63(6):819-830. doi: 10.1007/s40262-024-01375-2. Epub 2024 May 9. PMID 38722461